CLINICAL TRIAL: NCT02779140
Title: A Phase I, Double-Blind, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of NTM-1632 vs Placebo Administered Intravenously in Healthy Adults
Brief Title: Phase I, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of NTM-1632
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0024; HHSN272201300017I
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2017-04

CONDITIONS: Botulism
Keywords: BoNT; botulinum; Botulism; Clostridium; Neurotoxin; NTM-1632
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.033 mg/kg NTM-1632 (Experimental): N=6 administered 0.033 mg/kg NTM-1632 IV, N=2 administered placebo IV
  Interventions: Biological: NTM-1632; Other: Placebo
- 0.165 mg/kg NTM-1632 (Experimental): N=6 administered 0.165 mg/kg NTM-1632 IV, N=2 administered placebo IV
  Interventions: Biological: NTM-1632; Other: Placebo
- 0.33 mg/kg NTM-1632 (Experimental): N=6 administered 0.33 mg/kg NTM-1632 IV, N=2 administered placebo IV
  Interventions: Biological: NTM-1632; Other: Placebo

INTERVENTIONS:
Biological: NTM-1632 — Monoclonal antibody mixture of XB10, XB18, and XB23
Other: Placebo — Placebo

SUMMARY:
This is a Phase I, randomized, double-blind, placebo controlled dose escalation trial to evaluate NTM-1632 in three dose cohorts (A: 0.033 mg/kg, B: 0.165 mg/kg, and C: 0.33 mg/kg). NTM-1632 is a mixture of three monoclonal antibodies designed to treat botulinum neurotoxin BoNT/B poisoning in adults. Dose cohorts A, B, and C will be randomized 2:6, placebo:therapeutic, with a total study population of 24. The study duration is projected to be approximately 8 months, with subject participation in cohort A being approximately 13 weeks, and subject participation in cohort B and C being approximately 17 weeks. The primary objectives of this study are to assess the safety and tolerability of escalating doses of NTM-1632 administered intravenously in healthy adults.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo controlled dose escalation trial to evaluate NTM-1632 in three dose cohorts (A: 0.033 mg/kg, B: 0.165 mg/kg, and C: 0.33 mg/kg). NTM-1632 is a mixture of three monoclonal antibodies designed to treat botulinum neurotoxin BoNT/B poisoning in adults. Dose cohorts A, B, and C will be randomized 2:6, placebo:therapeutic, with a total study population of 24. The study duration is projected to be approximately 8 months, with subject participation in cohort A being approximately 13 weeks, and subject participation in cohort B and C being approximately 17weeks. The primary objectives of this study are to assess the safety and tolerability of escalating doses of NTM-1632 administered intravenously in healthy adults. The secondary objectives are to 1) assess the pharmacokinetic characteristics of NTM-1632 following a single intravenous administration and 2) assess the immunogenicity of NTM-1632 following a single intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed 2. Healthy male or healthy, non-pregnant, non-lactating female 3. Willingness to comply and be available for all protocol procedures including inpatient confinement for 36-48 hours 4. Age between 18 and 45 years, inclusive on the day of infusion 5. Body Mass Index (BMI) of >/=18.5 and </=30 kg/m2 6. If the subject is female and of childbearing potential, she has a negative serum pregnancy test at screening and negative urine test within 24 hours prior to infusion. Note: A woman is considered of childbearing potential unless post-menopausal (>/= 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation or successful Essure placement with documented confirmation test at least 3 months after the procedure. 7. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception, for up to visit 12 of the study. Note: Acceptable contraception methods are restricted to effective devices (Intrauterine Contraceptive Devices , NuvaRing®) or licensed hormonal products with use of method for a minimum of 28 days prior to dosing, condoms or diaphragm with spermicidal agents, monogamous relationship with a vasectomized partner. 8. The hemoglobin, platelet count, white blood cell count and absolute neutrophil count are within normal limits 9. The urine dipstick results on protein, glucose and blood are negative or trace. Note: Menstruating females failing inclusion criteria due to a positive blood on urine dipstick may be retested following cessation of menses. 10. Chemistry screening laboratory tests as outlined in Section 7.5.1.4 are in the normal reference range. Note: The following exceptions to laboratory normal reference ranges are allowed: Creatinine, Blood Urea Nitrogen (BUN), total bilirubin, AST, ALT, chloride, lipase, amylase, Prothrombin Time (PT), Partial Thromboplastin Time (PTT) below the lower limit of normal (LLN); CK less than 400mg/ml; Glucose, potassium, CO2, total protein, and alkaline phosphatase with a toxicity grade of 1 is allowable; Chlorides and albumin above the upper limit of normal (ULN). Laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once. Abnormalities in mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV), and nucleated red blood cell count (NRBC CT), which are included in a complete blood count with differential, will not be exclusions. 11. Has adequate venous access for the infusion 12. The urine drug screen is negative 13. Breathalyzer test is negative 14. Available for follow-up for the duration of the study. 15. Agrees not to participate in vigorous activity 72 hours prior to dosing through day 15 post dosing.

Exclusion Criteria:

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject. Note: Chronic medical conditions include diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; Coronary artery disease; Chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease (except previous asthma which has required no treatment for the past year); 2. History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins. Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema 3. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds) 4. Clinically significant abnormal electrocardiogram at screening. Note: Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator 5. Positive serology results for HIV, HBsAg, or HCV antibodies 6. Febrile illness with temperature >37.6°C within 7 days of dosing 7. Pregnant or breastfeeding 8. Donated blood within 56 days of enrollment 9. Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure 10. Treatment with another investigational drug within 28 days of dosing 11. Treatment with a monoclonal antibody at any time in the past 12. Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given 13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements 14. Use of H1 antihistamines or beta-blockers within 5 days of dosing 15. Use of any prohibited medication within 28 days prior to study entry or planned use during the study period Note: Prohibited medications include immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents; any vaccine (licensed or investigational) 16. Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin 17. Any previous injection or planned injection within 4 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason 18. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety 19. Plans to enroll or is already enrolled in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period. Note: Includes trials that have a study intervention such as a drug, biologic, or device 20. Is a study site employee or staff who are paid entirely or partially by the OCRR contract for the DMID-funded trial. Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators 21. Systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg 22. Resting heart rate <50 or >100 beats per minute 23. Oral temperature = 38°C (100.4°F)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
The occurrence of Adverse Events from administration of NTM-1632 | Day 1 to 57
The occurrence of changes from baseline in clinical safety laboratory values following administration of NTM-1632 | Screening, days -1, 2, 4, 8, 15, 29, 91
The occurrence of changes from baseline in ECG parameters post administration of NTM-1632 | Screening, day 1
The occurrence of changes from baseline in physical examination following administration of NTM-1632 | Screening, days -1, 1, 2
The occurrence of changes from baseline in vital signs following administration of NTM-1632 | Screening, days -1, 1, 2, 3, 4, 8, 15, 29, 43, 57, 91, 121
The occurrence of Serious Adverse Events following administration of NTM-1632 | Day 1 to 121

SECONDARY OUTCOMES:
The assessment of area-under-the-curve for concentration vs time (AUC(0-t)) for each of the three monoclonal antibodies of NTM-1632 | Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 91, 121
The assessment of maximum plasma titer/concentration (Cmax) for each of the three monoclonal antibodies of NTM-1632 | Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 91, 121
The assessment of time to maximum concentration (Tmax) for each of the three monoclonal antibodies of NTM-1632 | Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 91, 121
The presence of human anti-human antibodies in 0.165 mg/kg and 0.33 mg/kg dosing cohorts | Day 121
The presence of human anti-human antibodies in all dosing cohorts | Days -1, 1, 29, 57, 91

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Human Vaccine Institute - Duke Clinical Vaccine Unit, Durham, North Carolina, United States

REFERENCES:
- [Derived] Guptill JT, Raja SM, Juel VC, Walter EB, Cohen-Wolkowiez M, Hill H, Sendra E, Hauser B, Jackson P, Swamy GK. Safety, Tolerability, and Pharmacokinetics of NTM-1632, a Novel Mixture of Three Monoclonal Antibodies against Botulinum Toxin B. Antimicrob Agents Chemother. 2021 Jun 17;65(7):e0232920. doi: 10.1128/AAC.02329-20. Epub 2021 Jun 17. PMID 33875433